CLINICAL TRIAL: NCT05653869
Title: A Phase 1/1b Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of APS03118 in Adult Patients With Unresectable Locally Advanced or Metastatic Solid Tumors Harboring RET Mutations or Fusions
Brief Title: A Study of APS03118 in Advanced Solid Tumors Harboring RET Mutations or Fusions
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Applied Pharmaceutical Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APS-RET-102
Record Dates: First submitted 2022-11-15; First posted 2022-12-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: RET-altered Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APS03118 Dose Escalation (Experimental): APS03118 administered orally
  Interventions: Drug: APS03118

INTERVENTIONS:
Drug: APS03118 — Participant received APS03118 orally until evidence of unacceptable toxicity, progressed disease, consent withdrawal or with drawl from the study at the discretion of the investigator.
  Other Names: APS03118 administrated orally

SUMMARY:
This is a Phase 1/1b, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary antineoplastic activity of APS03118 administered orally in participants with RET-altered solid tumors.

DETAILED DESCRIPTION:
After being informed about the study procedure and potential risks and benefits, all patients giving written informed consent will undergo a 4-week screening period to determine eligibility for study entry. The eligible participants will be enrolled using a rolling 6 dose escalation scheme to identify MTD and/or RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older
2. Have histological or cytological confirmation of unresectable locally advanced or metastatic solid tumors harboring oncogenic RET mutations or fusions confirmed by NGS. Site may identify patients with a RET-mutated or RET-fusion solid tumor before the formal screening.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Resolution of all toxic effects of prior therapies to Grade 1 or below according to NCI CTCAE version 5.0 (except alopecia or Grade 2 neuropathy);
5. Patients with asymptomatic brain metastases if they have been previously treated, demonstrated no progression at least for 1 months before Screening, are asymptomatic and have had no requirement for steroids or enzyme inducing anticonvulsants in the last 14 days before Screening
6. Adequate organ function

Exclusion Criteria:

1. Have a locally advanced solid tumor that is a candidate for curative surgery treatment through radical surgery and/or radiotherapy.
2. Have an active fungal, bacterial, and/or active untreated viral infection
3. The patient has a serious pre-existing medical condition(s)
4. Have received or will receive a COVID-19 vaccine within 1 month before the first dose of APS03118.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs during Cycle 1 in dose-escalation cohorts | Within the 28 days of the first APS03118 dose for each patient
The maximum tolerated dose (MTD) and / or recommended Phase II dose (RP2D) | Approximately 15 months
  The MTD is defined as the maximum dose at which the incidence of dose-limiting toxicities (DLTs) during Cycle 1 is below 30%(<2/6)

SECONDARY OUTCOMES:
Adverse events(AE) | Approximately 24 months
Peak Plasma Concentration (Cmax) | Up to approximately 1 month
Area under the plasma concentration versus time curve (AUC) | Up to approximately 1 month
Time to Maximum Concentration (Tmax) | Up to approximately 1 month
Degree of accumulation | Up to approximately 1 month
Overall Response Rate (ORR) | Up to approximately 24 months
  As assessed by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Duration of response (DOR) | Up to approximately 24 months
Best of response (BOR) | Up to approximately 24 months
Disease Control Rate (DCR) | Up to approximately 24 months
Progress Free Survival (PFS) | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No